CLINICAL TRIAL: NCT02070991
Title: A Prospective, Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group, 12-week Study to Evaluate the Safety and Tolerability of Macitentan in Subjects With Combined Pre- and Post-capillary Pulmonary Hypertension (CpcPH) Due to Left Ventricular Dysfunction
Brief Title: Clinical Study to Evaluate the Safety and Tolerability of Macitentan in Subjects With Combined Pre- and Post-capillary Pulmonary Hypertension (CpcPH) Due to Left Ventricular Dysfunction
Acronym: MELODY-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-055G201
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Hypertension
Keywords: pre- and post-capillary pulmonary hypertension; CpcPH
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macitentan (Experimental): oral tablet, 10 mg once daily.
  Interventions: Drug: Macitentan
- Placebo (Placebo Comparator): Matching placebo, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macitentan — oral tablet, 10 mg once daily
  Other Names: ACT-064992
  Arms: Macitentan
Drug: Placebo — matching placebo
  Other Names: matching placebo
  Arms: Placebo

SUMMARY:
Study to evaluate if macitentan is safe and tolerable enough to be used for treatment of subjects with combined pre- and post-capillary pulmonary hypertension (CpcPH) due to left ventricular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females >=18 years of age
2. Subjects with combined pre-and post-capillary Pulmonary Hypertension (CpcPH) due to left ventricular dysfunction (subset of WHO groups 2.1 and 2.2)
3. Optimized diuretic therapy

Exclusion Criteria:

1. Types of Pulmonary Hypertension other than WHO groups 2.1 and 2.2 (Nice classification)
2. Administration of PAH-specific therapy (i.e., Endothelin receptor antagonists (ERAs), Prostanoids, Phosphodiesterase 5 (PDE-5) inhibitors, guanylate cyclase stimulators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Roux, PhD, Study Chair — Actelion
Locations (32):
- United States (6):
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan Internal Medicine Cardiology, Pulmonary Hypertension Program, Ann Arbor, Michigan
  - Washington University School of Medicine - Center for Advanced Med, St Louis, Missouri
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Houston Methodist Hospital - Heart Failure/Pulm Hypertension, Houston, Texas
- Austria (2):
  - Krankenhaus der Elisabethinen Linz, 2. Interne Abteilung, Linz
  - Medical University of Vienna and AKH Cardiology, Vienna
- Belgium (2):
  - Hôpital Erasme, Cliniques Universitaires de Bruxelles, Cardiologie, Brussels
  - University Hospital Gasthuisberg / Interne Geneeskunde - I.G. Pneumologie, Leuven
- Vancouver General Hospital - The Lung, Vancouver, Canada
- Czechia (4):
  - FN Brno-Bohunice, I. interní kardiologická klinika, Brno
  - FN Olomouc, 1. Interní klinika - kardiologická, Olomouc
  - IKEM (Institut klinické a experimentální medicíny, Institute for Clinical and Experimental Medicine), Prague
  - Lékařská fakulta a Všeobecná fakultní nemocnice v Praze, II. Interní klinika kardiologie a angiologie, Prague
- Hôpital Charles Nicolle Service de Cardiologie, Rouen, France
- Germany (4):
  - DRK Klinken Berlin Kopenick Klinik für Innere Medizin Kardiologie, Berlin
  - Universitätsklinikum Köln Herzzentrum / Klinik III für Innere Medizin (Kardiologie, Pneumologie, Angiologie und Intensivmedizin), Cologne
  - Universitätsklinik Schleswig-Holstein Campus Kiel Klinik für Innere Medizin III Kardiologie und Angiologie, Kiel
  - Klinikum der Universität München Medizinische Klinik und Poliklinik 1 - Großhadern Schwerpunkt Pneumologie, Munich
- Israel (4):
  - Carmel Medical Center, Pulmonary Unit, Haifa
  - Institute of Pulmonology Hadassah Medical Centre : Ein Karem, Jerusalem
  - Kaplan Medical Centre / Pulmonary Institute and Department of Medicine, Rehovot
  - The Chaim Sheba Medical Center / The Institute of Pulmonology, Physiology and Exercise, Tel Litwinsky
- Italy (2):
  - A.O. Universitaria Policlinico S. Orsola-Malpighi - Dipartimento di Medicina Specialistica, Diagnostica e Sperimentale - Unità Operativa di Cardiologia, Bologna
  - Ospedali Riuniti Di Trieste, Trieste
- Spain (4):
  - Hospital Vall d´Hebron Servicio de Cardiologia, Barcelona
  - Hospital Clinic Servicio de Cardiologia, Barcelona
  - Hospital Reina Sofia Servicio de Cardiologia, Córdoba
  - Hospital Universitario 12 Octubre Servicio de Cardiología, Madrid
- Switzerland (2):
  - Universitätsklinik für Kardiologie Schweizer Herz- und Gefässzentrum Bern, Bern
  - Centre Hospitalier Universitaire Vaudois Service de Cardiologie, Lausanne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened from 28 sites across Europe and North America in 11 countries (Austria, Belgium, Canada, Czech Republic, Germany, France, Israel, Italy, Spain, Switzerland, USA).
Pre-assignment Details: Of the 88 participants screened 63 were randomized in a 1:1 ratio to macitentan 10 mg (N = 31) or placebo (N = 32).
Groups:
- Macitentan: Macitentan 10 mg to be taken once daily, oral use, film-coated tablet
- Placebo: Matching placebo to be taken once daily, oral use, film-coated tablet
Period: Overall Study
Arm/Group | Macitentan | Placebo
Started | 31 | 32
Completed | 28 | 32
Not Completed | 3 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 70.0 [67.0 to 73.0] | 72.0 [68.0 to 75.5] | 71.0 [67.0 to 75.0]
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 5 | 3 | 8
  65-84 years | 26 | 28 | 54
  ≥ 85 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 6 | 16 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 30 | 31 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 1 | 1
  American Indian or Alaska Native | 1 | 0 | 1
  White | 30 | 30 | 60
  Other | 0 | 1 | 1
Time from Left Ventricular Dysfunction (LVD) diagnosis [Median (Inter-Quartile Range); unit: years] | 0.9 [0.1 to 5.4] | 1.5 [0.4 to 3.4] | 1.3 [0.2 to 4.2]
Time from Combined pre- and post-capillary Pulmonary Hypertension (CpcPH) diagnosis [Median (Inter-Quartile Range); unit: years] — Population: The value of 1 patient is missing in the macitentan group.
  years
    number analyzed (Participants) | 30 | 32 | 62
    (all) | 0.2 [0.0 to 1.4] | 0.2 [0.0 to 0.5] | 0.2 [0.0 to 0.5]
New York Heart Association (NYHA) Functional Class at baseline [Count of Participants; unit: Participants] — Class I: No symptoms and no limitation in ordinary physical activity, e.g., shortness of breath when walking, climbing stairs etc. Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. Class III: Marked limitation in activity due to symptoms, even during less-than ordinary activity, e.g., walking short distances (20-100 m). Comfortable only at rest. Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    Class I | 0 | 0 | 0
    Class II | 5 | 10 | 15
    Class III | 26 | 22 | 48
    Class IV | 0 | 0 | 0
6-minute walk distance (6MWD) at baseline [Median (Inter-Quartile Range); unit: meter] | 300.0 [216.0 to 435.0] | 305.0 [206.5 to 379.5] | 300.0 [215.0 to 410.0]
Participants with Atrial Fibrillation at baseline [Count of Participants; unit: Participants]
  Yes | 22 | 24 | 46
  No | 9 | 8 | 17
Participants with Diabetes Mellitus Type II [Count of Participants; unit: Participants]
  Yes | 14 | 13 | 27
  No | 17 | 19 | 36
Participants with Right Heart Failure (RHF) [Count of Participants; unit: Participants]
  Yes | 7 | 11 | 18
  No | 24 | 21 | 45
Participants with Systemic Hypertension [Count of Participants; unit: Participants]
  Yes | 30 | 27 | 57
  No | 1 | 5 | 6
Participants with Chronic Kidney Disease (CKD) [Count of Participants; unit: Participants]
  Yes | 8 | 6 | 14
  No | 23 | 26 | 49
Left Ventricular Ejection Fraction (LEVF) at baseline as measured by Investigator [Count of Participants; unit: Participants]
  < 50% | 6 | 9 | 15
  ≥ 50% | 25 | 23 | 48
Pulmonary Vascular Resistance (PVR) at baseline [Median (Inter-Quartile Range); unit: dyn*sec/cm^5] | 450.0 [296.0 to 590.0] | 483.5 [362.0 to 738.5] | 462.0 [341.0 to 695.0]
Body Mass Index (BMI) at baseline [Median (Inter-Quartile Range); unit: kg/m^2] | 33.30 [28.80 to 38.30] | 31.15 [27.60 to 34.45] | 32.40 [28.70 to 36.00]
Participants with obesity (BMI > 30 kg/m^2) [Count of Participants; unit: Participants]
  Yes | 20 | 20 | 40
  No | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Significant Fluid Retention or Worsening in NYHA Functional Class (FC) up to End-of-treatment
Description: The main endpoint is the number of participants who had at least one of the following: A) significant fluid retention, defined as increase in body weight at any time by ≥ 5% or ≥ 5 kg from baseline due to fluid overload and/or parenteral administration of diuretics. B) Worsening of NYHA functional class from baseline.
Time Frame: From randomization up to End-of-Study (Week 12 + 30 days follow-up) plus 1 calendar day
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 31 | 32
Participants
  Total participants with at least one condition | 7 | 4
  Participants with fluid retention | 7 | 3
  Participants with worsening in NYHA FC | 1 | 2
  Participants with both conditions | 1 | 1
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; p = 0.3372, Fisher Exact; Difference between maci. and placebo = 10.08, 95% CI 2-sided [-15.07 to 33.26]

2. Secondary Outcome: NT-proBNP at Week 12 Expressed as Percent of Baseline NT-proBNP at Rest
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 6 patients are missing in both the macitentan and the placebo group.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline NT-proBNP
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 25 | 26
percentage of baseline NT-proBNP | 91.56 [72.37 to 115.83] | 118.90 [92.53 to 152.78]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (ratio of geom. means) = 0.77, 95% CI 2-sided [0.55 to 1.08]

3. Secondary Outcome: PVR at Rest at Week 12 Expressed as Percent of Baseline PVR at Rest
Description: Pulmonary vascular resistance (PVR) was assessed at rest by right heart catheterization (RHC).
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 11 patients in the macitentan group and of 8 patients in the placebo group are missing.
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of baseline PVR
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 20 | 24
percentage of baseline PVR | 66.31 [56.15 to 78.30] | 71.23 [51.35 to 98.81]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (ratio of geom. means) = 0.93, 95% CI 2-sided [0.64 to 1.36]

4. Secondary Outcome: Change From Baseline to Week 12 in Mean Pulmonary Arterial Pressure (mPAP)
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 10 patients in the macitentan group and of 7 patients in the placebo group are missing.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 21 | 25
mmHg
  mPAP at baseline | 44.6 [40.7 to 48.6] | 45.9 [41.7 to 50.1]
  mPAP at Week 12 | 41.1 [36.2 to 46.0] | 42.1 [37.5 to 46.7]
  Change in mPAP from baseline to Week 12 | -3.5 [-6.1 to -0.9] | -3.8 [-7.5 to -0.1]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (mean change from BL) = 0.3, 95% CI 2-sided [-4.3 to 4.9]

5. Secondary Outcome: Change From Baseline to Week 12 in Mean Right Atrial Pressure (mRAP)
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 10 patients in the macitentan group and of 7 patients in the placebo group are missing.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 21 | 25
mmHg
  mRAP at baseline | 12.1 [10.0 to 14.3] | 13.0 [11.0 to 14.9]
  mRAP at Week 12 | 11.2 [8.7 to 13.8] | 11.3 [9.2 to 13.5]
  Change in mRAP from baseline to Week 12 | -0.9 [-3.5 to 1.7] | -1.6 [-3.3 to 0.0]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (mean change from BL) = 0.7, 95% CI 2-sided [-2.2 to 3.6]

6. Secondary Outcome: Change From Baseline to Week 12 in Pulmonary Artery Wedge Pressure (PAWP)
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 11 patients in the macitentan group and of 8 patients in the placebo group are missing.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 20 | 24
mmHg
  PAWP at baseline | 19.1 [17.4 to 20.7] | 19.7 [18.2 to 21.2]
  PAWP at Week 12 | 19.9 [16.6 to 23.1] | 20.8 [17.8 to 23.7]
  Change in PAWP from baseline to Week 12 | 0.8 [-2.3 to 3.9] | 1.1 [-1.6 to 3.8]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (mean change from BL) = -0.3, 95% CI 2-sided [-4.2 to 3.7]

7. Secondary Outcome: Change From Baseline to Week 12 in Cardiac Index (CI)
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 11 patients in the macitentan group and of 8 patients in the placebo group are missing.
Measure: Mean (95% Confidence Interval); unit: L/min/m^2
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 20 | 24
L/min/m^2
  CI at baseline | 2.32 [2.02 to 2.61] | 2.33 [2.09 to 2.57]
  CI at Week 12 | 2.69 [2.36 to 3.02] | 2.30 [2.03 to 2.57]
  Change in CI from baseline to Week 12 | 0.37 [0.14 to 0.60] | -0.03 [-0.22 to 0.16]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (mean change from BL) = 0.40, 95% CI 2-sided [0.11 to 0.69]

8. Secondary Outcome: Change From Baseline to Week 12 in Diastolic Pulmonary Vascular Pressure Gradient (DPG)
Time Frame: From randomization up to end of treatment period (Week 12)
Population: The values of 11 patients in the macitentan group and of 8 patients in the placebo group are missing.
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Macitentan | Placebo
Number analyzed (Participants) | 20 | 24
mmHg
  DPG at baseline | 11.8 [9.0 to 14.5] | 11.4 [9.5 to 13.2]
  DPG at Week 12 | 7.0 [4.2 to 9.8] | 7.0 [3.7 to 10.4]
  Change in DPG from baseline to Week 12 | -4.8 [-7.2 to -2.3] | -4.3 [-7.5 to -1.1]
Statistical Analysis 1: Comparison: Macitentan vs Placebo; Test type: Superiority or Other; Treatment effect (mean change from BL) = -0.4, 95% CI 2-sided [-4.5 to 3.6]

ADVERSE EVENTS:
Time Frame: From study treatment initiation up to 30 days after study treatment discontinuation (Week 12 + 30 days)
Arm/Group | Macitentan | Placebo
All-Cause Mortality (participants affected / at risk) | 2/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 11/31 | 6/32
Other Adverse Events (participants affected / at risk) | 16/31 | 15/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=31) | Placebo (N=32)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=31) | Placebo (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 3 (3)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2) | 0 (0)
Walking distance test abnormal (Investigations) | 0 (0) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.